CLINICAL TRIAL: NCT02406469
Title: Comparative Effects of Milk With A2 Type Beta Casein Versus Milk With A1 and A2 Beta Casein Proteins on Gastrointestinal Physiology, Symptoms and Cognitive Behavior for the Health People Who Are Intolerant to Traditional Cow Milk
Brief Title: Effects Comparison of A1 and A2 Milk on Gastrointestinal Physiology, Symptoms and Cognitive Behavior
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: a2 Milk Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 14-SC-07-A2-01
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A1-A2 (Experimental): Oral consumption of milk containing both A1 and A2 type beta casein in intervention phase 1 and milk containing only A2 type beta casein in intervention phase 2.
  Interventions: Dietary Supplement: Oral consumption milk Tetra Pak
- Sequence A2-A1 (Placebo Comparator): Oral consumption of milk containing only A2 type beta casein in intervention phase 1 and milk containing both A1 and A2 type beta casein in intervention phase 2.
  Interventions: Dietary Supplement: Oral consumption milk Tetra Pak

INTERVENTIONS:
Dietary Supplement: Oral consumption milk Tetra Pak — Oral consumption of assigned products in the form of Tetra Pak (A1 or A2 milk according to randomization), 250 ml/time, 2 times daily after meal, for a total of 28 days (14 days in each intervention phase).

SUMMARY:
This is a single-site, double-blinded, randomized, controlled, 2X2 cross-over study aiming to compare effects of milk containing only A2 type beta casein versus milk containing both A1 and A2 beta casein proteins on the gastrointestinal physiology, symptoms and cognitive behaviour for the health people who are intolerant to traditional cow's milk.

DETAILED DESCRIPTION:
This is a single-site, double-blinded, randomized, controlled, cross-over study in healthy milk drinkers of 4 weeks' consumption with milk containing only A2 type beta casein (called A2 milk) versus milk containing both A1 and A2 beta casein proteins (called A1 milk) to compare the effects on gut inflammation (CRP, HB, IL-4, IgG, IgE, IgG1, IgG2a), gastrointestinal symptoms (via VAS score including Bloating, Abdominal pain, Flatulence, Break wind, Borborygmi), regional gut transit times (via 'Smart Pill') and behavioral well-being (CNAQ), and stool habits.

The cross-over study will take 2 phases (2 weeks in each phase) of product intervention, 2 weeks of wash-out before each intervention phase and then followed by 5 wks of statistical analysis and clinical report completed.

According to ICH-GCP Guidelines and Chinese regulations issued by SFDA, all subjects will be informed of study procedures and sign the informed consent before enrollment. At screening phase, subjects will be informed about study requirements, procedures, potential risks and benefits of participation. Subjects will not be enrolled into the study until ICF is well informed and accepted.

At the Screening phase, 100 subjects had the Urine galactose (U-gal) test to screen 45 subjects eligible for the study and they should simultaneously meet the Inclusion and Exclusion criteria. Subjects should be fasting on the morning of testing, and then drink 300 ml full-fat milk within 3-5 minutes. Empty the urine 1 hour after drinking, and collect midstream urine 2 hours after milk-consumption for urinary galactose test with symptom scores recorded accordingly. Urine galactose (U-gal) tests positive indicating the lactase deficiency, if it is accompanied by abdominal distension, abdominal pain and other symptoms of more than 1 item; it is identified as lactose intolerance.

100 subjects took part in the screening by U-gal test and forty-five (45) qualified subjects (stratified by male to female approximate ratio 1:1) will be enrolled into the study with assumed 11.1% attrition rate to keep 20 subjects per group to complete the cross-over study. Subjects will be enrolled in the study site authorized by Xin Hua Hospital during the screening phase. Sun Jianqin, Professor, leading PI, is responsible for the academic guidance to define all qualified subjects. The study will be conducted by the team of PIs and monitored by SPRIM CHINA in accordance with Chinese Good Clinical Practices (CGCP's). Subjects will sign the informed consent form before study intervention. Eligible subjects will be randomized into 2 groups, and one of two possible products sequences will be assigned, A1 milk or A2 milk. Subjects completed 2 weeks A1 or A2 intervention after initial 2 weeks of washout, and then cross over to the opposite intervention for 2 weeks after second 2 weeks of washout. The efficacy of the study products was evaluated by biomarkers in the blood or feces and linked questionnaires at the duration of the cross-over study.

During the study intervention, subjects need to visit the site every week; follow-up telephone will be made at the duration of wash-out phase and the related information will be collected by CRAs accordingly.

ELIGIBILITY:
Inclusion Criteria:

* 25~3568 years old male or female subjects who:
* Non-regular milk drinker with self-reported intolerance to commercial milk;
* Suffered from mild to moderate digestive discomfort after milk consumption;
* Have normal electrocardiograms (ECG) and blood pressure during quiet respiration;
* Agree not to take any medication, supplements, nutrition or other dairy products including acidophilus milk;
* Be willing to comply with all the requirements and procedures of the study;
* Agree to sign the informed consent form;
* Agree not to enroll in another interventional clinical research study while participating in this study;
* Fully understand the nature, objective, benefit and the potential risks and side effects of the study.

Exclusion Criteria:

* Female on pregnant or feeding；
* Have known dairy allergy;
* Have severe response to milk intolerance;
* Have history of faecal impaction;
* Trying to lose weight by following a diet or exercise regimen designed for weight loss, or taking any drug influencing appetite and any drug for weight loss for the last three months ;
* Have participated in similar dairy or probiotics-containing product's clinical trials within 3 months before the screening;
* Currently taking medicines for cardiovascular or metabolic disease;
* Have history of or be diagnosed of any of the following diseases that may affect the study results: gastrointestinal disorders, hepatopathy, nephropathy, endocrine disease, blood disorders, respiratory and cardiovascular diseases;
* Current or previous alcohol abuser, currently taking or took illicit drugs, substance or OTC prescription drugs in regular frequency which may affect gastrointestinal disorders and study result;
* Currently suffering from any gastrointestinal disorders or gastrointestinal disease, including but not limited to: irritable bowel syndrome, colitis, ulcerative colitis, celiac disease, irritable bowel syndrome(IBS);
* Had hospitalizations within 3 months before screening;
* Currently drug frequency user of that may affect the gastrointestinal function or immune system. As judged by investigator.

Ages: 25 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Serum levels of immune response markers in correlation to symptoms of intolerance | Baseline 1 (Day 0), end of intervention phase 1 (Day 14), baseline 2 (Day 28), end of intervention phase 2 (Day 42)
  Serum levels of interlukin-4, IgE, IgG1 and IgG2A

SECONDARY OUTCOMES:
Regional gut transit time | End of intervention phase 1 (Day 14), end of intervention phase 2 (Day 42)
  Measurement using "Smart Pill" device
Fecal short chain fatty acid measurements | Baseline 1 (Day 0), end of intervention phase 1 (Day 14), baseline 2 (Day 28), end of intervention phase 2 (Day 42)
  Markers for absorption of nutrients and gut inflammation
Gastrointestinal symptoms (VAS score) | Daily from Day 0 to Day 42
  Evaluated through VAS score reporting
Stool frequency | Daily from Day 0 to Day 42
Stool consistency (Bristol Score) | Daily from Day 0 to Day 42
  Measured via Bristol Score
Response time and error rate | Baseline 1 (Day 0), end of intervention phase 1 (Day 14), baseline 2 (Day 28), end of intervention phase 2 (Day 42)
  Markers for change of cognition function evaluated via Subtle Cognitive Impairment Test (SCIT)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Clarke, PhD, Study Director — a2 Milk Company Ltd.

REFERENCES:
- [Derived] Deth R, Clarke A, Ni J, Trivedi M. Clinical evaluation of glutathione concentrations after consumption of milk containing different subtypes of beta-casein: results from a randomized, cross-over clinical trial. Nutr J. 2016 Sep 29;15(1):82. doi: 10.1186/s12937-016-0201-x. PMID 27680716
- [Derived] Jianqin S, Leiming X, Lu X, Yelland GW, Ni J, Clarke AJ. Effects of milk containing only A2 beta casein versus milk containing both A1 and A2 beta casein proteins on gastrointestinal physiology, symptoms of discomfort, and cognitive behavior of people with self-reported intolerance to traditional cows' milk. Nutr J. 2016 Apr 2;15:35. doi: 10.1186/s12937-016-0147-z. PMID 27039383